CLINICAL TRIAL: NCT00998192
Title: A Phase 2 Study of Intravenous Administration of REOLYSIN® (Reovirus Type 3 Dearing) in Combination With Paclitaxel and Carboplatin in Patients With Squamous Cell Carcinoma of the Lung
Brief Title: A Study of REOLYSIN® in Combination With Paclitaxel and Carboplatin in Patients With Squamous Cell Carcinoma of the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncolytics Biotech (Industry)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REO 021
Record Dates: First submitted 2009-10-15; First posted 2009-10-20 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2015-08

CONDITIONS: Metastatic or Recurrent Squamous Cell Carcinoma of the Lung
Keywords: carcinoma; squamous cell; lung; REOLYSIN; chemotherapy; carboplatin; paclitaxel; Carcinoma, Squamous Cell of the Lung
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma | interventions — reolysin; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: REOLYSIN — 3x10E10 TCID50 1 hour intravenous infusion, administered on Days 1,2,3,4,and 5 of a 21-day cycle
Drug: Paclitaxel — 200 mg/m2, 3-hour intravenous infusion, given on Day 1 of a 21-day cycle
  Other Names: Taxol
Drug: Carboplatin — 6 AUC mg/mL min, 30-min intravenous infusion, given on Day 1 of a 21-day cycle
  Other Names: Paraplatin

SUMMARY:
The purpose of this Phase 2 study is to investigate whether intravenous administration of REOLYSIN therapeutic reovirus in combination with paclitaxel and carboplatin is effective and safe in the treatment of squamous cell carinoma of the lung.

DETAILED DESCRIPTION:
Lung cancer remains the most common cancer and cause of cancer-related mortality in the United States. In 2008, there was an estimated 215,000 new cases of lung cancer diagnosed and roughly 162,000 deaths from lung cancer (NCI 2009). The majority (85%) of patients with a diagnosis of lung cancer will have non-small cell lung cancer (NSCLC).

The combination of paclitaxel and carboplatin has become the most commonly prescribed chemotherapy regimen for the treatment of advanced NSCLC in the United States. Laboratory studies of combinations of REOLYSIN with a variety of chemotherapeutic agents has shown that the combination of REOLYSIN and paclitaxel was invariably synergistic, even in cells with drug resistance or limited sensitivity to the reovirus. Moreover, reovirus activity was dramatically increased in the presence of the taxane.

The Phase 2 study is designed to characterize the efficacy and safety of REOLYSIN given intravenously in combination with paclitaxel and carboplatin every 3 weeks in patients with squamous cell carinoma of the lung.

Response is a primary endpoint of this trial.

The safety of the treatment combination will be assessed by the evaluation of the type, frequency and severity of adverse events, changes in clinical laboratory tests, immunogenicity and physical examination.

Patients may continue to receive chemotherapy combined with REOLYSIN for up to 8 cycles and may continue indefinitely on REOLYSIN monotherapy under this protocol, provided they have not experienced either progressive disease or unacceptable drug-related toxicity that does not respond to either supportive care or dose reduction.

ELIGIBILITY:
Inclusion Criteria:

* have histologically or cytologically confirmed metastatic stage IIIB (pleural effusion; IVA on revised IASLC staging) or stage IV, or recurrent squamous cell carcinoma of the lung.
* have measurable disease.
* be chemotherapy naïve for their metastatic or recurrent SCCLC, with some exceptions.
* have NO continuing acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedures.
* have an ECOG Performance Score of ≤ 2.
* have a life expectancy of at least 3 months.
* absolute neutrophil count (ANC) ≥ 1.5 x 10^9; Platelets ≥ 100 x10^9 (without platelet transfusion);Hemoglobin ≥ 9.0 g/dL (with or without RBC transfusion); Serum creatinine ≤ 1.5 x upper limit of normal (ULN); Bilirubin ≤ 1.5 x ULN; AST/ALT ≤ 2.5 x ULN.
* negative pregnancy test for females with childbearing potential.

Exclusion Criteria:

* receive concurrent therapy with any other investigational anticancer agent while on study.
* have a known past or current history of brain metastasis(es).
* be on immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* be a pregnant or breast-feeding woman.
* have clinically significant cardiac disease.
* have dementia or altered mental status that would prohibit informed consent.
* have any other acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate (complete response (CR) + partial response (PR)) of the treatment regimen in the study population | 6 months

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of the treatment regimen in the study population as measured by adverse events associated with the study treatment, and defined by established criteria. | Within 30 days of last dose of REOLYSIN
To assess progression-free survival (PFS) for the treatment regimen in the study population. | 9-12 months
Determine the proportion of patients receiving the treatment who are alive and free of disease progression at 6 months. | 6 months
To determine overall survival with the treatment regimen in the study population | 9-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alain Mita, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (17):
- United States (17):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Ocala Oncology Center, Ocala, Florida
  - Illinois Cancer Specialists, Niles, Illinois
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Advanced Oncology Associates, Armonk, New York
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Medical Oncology Associates of Wyoming Valley, Kingston, Pennsylvania
  - Texas Oncology - Arlington South, Arlington, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Texas Oncology - Garland, Garland, Texas
  - Texas Oncology - Lewisville, Lewisville, Texas
  - Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Lynchburg Hematology Oncology Clinic, Lynchburg, Virginia